CLINICAL TRIAL: NCT04086147
Title: Chinese Acute Tissue-based Imaging Selection for Lysis in Stroke: a Prospective, Multicentre, Randomized, Open-label, Rater-blinded, Randomized Trial
Brief Title: CHinese Acute Tissue-Based Imaging Selection for Lysis In Stroke -Tenecteplase
Acronym: CHABLIS-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: The First Affiliated Hospital of Shanxi Medical University (Other); Ningbo No. 1 Hospital (Other); Zhejiang Province People's Hospital (Unknown); Shanghai 5th People's Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai 6th People's Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); The Second People's Hospital of Huai'an (Other); Pu'er City People's Hospital (Unknown); ShuGuang Hospital (Other); Shanghai East Hospital (Other); First People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Qiang Dong, Director of Neurology Department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017YFC1308201
Record Dates: First submitted 2019-04-15; First posted 2019-09-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: acute ischemic stroke; large vessel occlusion; thrombolysis; tenecteplase; dosage; computed tomography; magnetic resonance imaging; diffusion weighted imaging; early combined imaging outcomes; modified Rankin scale; time window beyond 4.5 hours
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose tenecteplase (Experimental)
  Interventions: Drug: Low dose tenecteplase
- High dose tenecteplase (Experimental)
  Interventions: Drug: High dose tenecteplase

INTERVENTIONS:
Drug: Low dose tenecteplase — Intravenous (IV) tenecteplase 0.25 mg/kg (single bolus; maximum dose 25 mg)
  Arms: Low dose tenecteplase
Drug: High dose tenecteplase — Intravenous (IV) tenecteplase 0.32 mg/kg (single bolus; maximum dose 32 mg)
  Arms: High dose tenecteplase

SUMMARY:
To select the best dosage of tenecteplase for acute ischemic stroke patients (onset time 4.5-24h) of large vessel occlusion using early combined CT/MR imaging outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with anterior circulation acute ischaemic stroke
2. Time from onset to treatment 4.5h-24h
3. Patient's age is ≥18 years
4. Pre-stroke mRS score of <= 2
5. Clinically significant acute neurologic deficit
6. Vessel occlusion or severe stenosis ( ICA, MCA-M1/M2, ACA) on computed tomography angiography (CTA)/MRA
7. Multimodal CT/magnetic resonance imaging: perfusion lesion volume (DT > 3 s) to infarct core volume ratio (rCBF<30% or diffusion-weighted imaging lesion) >1.2, absolute difference >10 ml, and ischemic core volume <70ml
8. Informed consent was obtained from patients.

Exclusion Criteria:

1. Intracranial hemorrhage or subarachnoid hemorrhage identified by CT or MRI
2. Rapidly improving symptoms (patient with an NIHSS score decrease to < 4 at randomization)
3. Pre-stroke mRS score of > 2
4. Contraindication to imaging with CT/magnetic resonance imaging with contrast agents
5. Infarct core >1/3 middle cerebral artery (MCA) territory
6. Platelet count < 100x10^9/L
7. Symptoms were caused by low blood glucose < 2.7 mmol/l
8. Severe uncontrolled hypertension, i.e. systolic blood pressure >= 180 mmHg or diastolic blood pressure >=100 mmHg
9. Current use of warfarin with a prolonged prothrombin time (INR > 1.7 or prothrombin time > 15s)
10. Use of low molecular weight heparin within 24 hours
11. Use of non-vitamin K antagonist oral anticoagulants (NOACs) within 48 hours
12. Use of glycoprotein IIb - IIIa inhibitors within 72 hours.
13. Arterial puncture at noncompressible site in previous 7 days
14. Major surgery in previous 14 days which poses risk in the opinion of the investigator
15. Recent gastrointestinal or urinary tract hemorrhage (within previous 21 days)
16. Significant head trauma or prior stroke in previous 3 months
17. History of previous intracranial hemorrhage, intracranial neoplasm, arteriovenous malformation, or aneurysm. Risks were considered by the investigator
18. Hereditary or acquired haemorrhagic diathesis
19. Active internal bleeding
20. Symptoms suggestive or recent acute pancreatitis, active gastrointestinal ulcer
21. Severe liver disease, including liver failure, cirrhosis, portal hypertension and active hepatitis
22. Pregnancy
23. Various dying diseases with life expectancy ≤3 months
24. Other conditions in which doctors believe that participating in this study may be harmful to the patient
25. Patients participated in any observational trial in 30 days
26. Allergic to the test drug and its ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Favourable outcome: patients without endovascular therapy obtained >50% reperfusion at 4-6 hours | 4-6 hours
  Without endovascular therapy: >50% reperfusion on computed tomography perfusion (CTP) at 4-6 hours
Favourable outcome: patients with endovascular therapy: mTICI score 2b or better at initial angiogram | Before endovascular therapy
  With endovascular therapy: mTICI score 2b or better at initial angiogram after thrombolysis before endovascular therapy
Favourable outcome: no symptomatic intracranial hemorrhage at 24-36 hours | 24-36 hours
  No symptomatic intracranial hemorrhage at 24-36 hours

SECONDARY OUTCOMES:
Imaging efficacy outcome: recanalization rate on CT/magnetic resonance angiography | 4-6 hours
  Recanalization rate on CTA/MRA at 4-6 hours
Imaging efficacy outcome: Infarct volume growth (ml) at 3-5 days on MRI | 3-5 days
  Infarct volume growth (ml) at 3-5 days on MRI
Clinical efficacy outcome: major neurological improvement at 24-36 hours ( NIHSS reduction ≥8 or return to 0-1) | 24-36 hours
  Major neurological improvement at 24-36 hours ( NIHSS reduction >8 or return to 0-1)
Clinical efficacy outcome: NIHSS change | 24-36 hours
  NIHSS change at 24-36 hours as a continuous variable
Clinical efficacy outcome: excellent functional outcome (modified Rankin scale 0-1) vs (modified Rankin scale 2-6) at 90 days | 90 days
  Excellent functional outcome (modified Rankin scale 0-1) vs (modified Rankin scale 2-6) at 90 days. The modified Rankin Scale is a simple 7-point assessment that includes reference to both limitations in activity and changes in lifestyle. 0=No symptoms at all; no limitations and no symptoms. 1=No significant disability despite symptoms; able to carry out all usual duties and activities. 2=Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance. 3=Moderate disability; requiring some help, but able to walk without assistance. 4=Moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance. 5=Severe disability: bedridden, incontinent, and requiring constant nursing care and attention. 6=Death.
Clinical efficacy outcome: good functional outcome (modified Rankin scale 0-2) vs (modified Rankin scale 3-6) at 90 days | 90 days
  Good functional outcome (modified Rankin scale 0-2) vs (modified Rankin scale 3-6) at 90 days. The modified Rankin Scale is a simple 7-point assessment that includes reference to both limitations in activity and changes in lifestyle. 0=No symptoms at all; no limitations and no symptoms. 1=No significant disability despite symptoms; able to carry out all usual duties and activities. 2=Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance. 3=Moderate disability; requiring some help, but able to walk without assistance. 4=Moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance. 5=Severe disability: bedridden, incontinent, and requiring constant nursing care and attention. 6=Death.
Clinical efficacy outcome: modified Rankin scale shift | 90 days
  Modified Rankin scale shift at 90 days. The modified Rankin Scale is a simple 7-point assessment that includes reference to both limitations in activity and changes in lifestyle. 0=No symptoms at all; no limitations and no symptoms. 1=No significant disability despite symptoms; able to carry out all usual duties and activities. 2=Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance. 3=Moderate disability; requiring some help, but able to walk without assistance. 4=Moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance. 5=Severe disability: bedridden, incontinent, and requiring constant nursing care and attention. 6=Death.
Imaging safety outcome: Intracranial hemorrhage of any volume at 24-36 hours | 24-36 hours
  Intracranial hemorrhage of any volume at 24-36 hours
Imaging safety outcome: parenchymal hematoma 2 at 24-36 hours | 24-36 hours
  Parenchymal hematoma 2 at 24-36 hours
Imaging safety outcome: Symptomatic intracranial hemorrhage at 24-36 hours | 24-36 hours
  Symptomatic intracranial hemorrhage at 24-36 hours
Clinical safety outcome: Poor functional outcome (mRS 5, 6) at 90 days | 90 days
  Poor functional outcome (mRS 5, 6) at 90 days. The modified Rankin Scale is a simple 7-point assessment that includes reference to both limitations in activity and changes in lifestyle. 0=No symptoms at all; no limitations and no symptoms. 1=No significant disability despite symptoms; able to carry out all usual duties and activities. 2=Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance. 3=Moderate disability; requiring some help, but able to walk without assistance. 4=Moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance. 5=Severe disability: bedridden, incontinent, and requiring constant nursing care and attention. 6=Death.
Clinical safety outcome: Rate of systemic bleeding | 24 hours
  Rate of systemic bleeding within 24 hours
Barthel index | 90 days
  Barthel index at 90 days. The Barthel Index is a scale that indicates the ability to perform a selection of activities of daily living. It comprises 10 items (tasks), with total scores ranging from 0 (worst mobility in activities of daily living) to 100 (full mobility in activities of daily living) and it has adequate clinimetric (quality of clinical measurements) properties in stroke rehabilitation. In the index, the 10 items have these scoring combinations: a) 0 and 5, b) 0, 5 and 10, or c) 0, 5, 10 and 15. These items in the Barthel Index address a patient's ability in feeding, bathing, grooming, dressing, bowel and bladder control, toileting, chair transfer, ambulation and stair climbing.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu X, Hong L, Zhao G, He Z, Wang X, Zhu J, Li S, Zhang A, Cao N, Ling Y, Chen X, Guo Y, Fang Q, Wang Z, Dong Q, Cheng X. Regional perfusion parameters as potential indicators of parenchymal hematoma risk following reperfusion therapy for acute ischemic stroke in the extended time window. Ther Adv Neurol Disord. 2025 Dec 21;18:17562864251406032. doi: 10.1177/17562864251406032. eCollection 2025. PMID 41446320
- [Derived] Hong L, Zhu J, He Z, Wang X, Li S, Liu X, Ling Y, Yang L, Fang Q, Dong Q, Cheng X; CHABLIS-T Investigators. Effect of Time Delay on Reperfusion After Tenecteplase in an Extended Time Window: Analysis From the CHABLIS-T Trials. J Am Heart Assoc. 2025 Jun 17;14(12):e040994. doi: 10.1161/JAHA.124.040994. Epub 2025 Jun 11. PMID 40497495
- [Derived] Cheng X, Hong L, Churilov L, Lin L, Ling Y, Zhang J, Yang J, Geng Y, Wu D, Liu X, Zhou X, Zhao Y, Zhai Q, Zhao L, Chen Y, Guo Y, Yu X, Gong F, Sui Y, Li G, Yang L, Gu HQ, Wang Y, Parsons M, Dong Q; CHABLIS-T collaborators. Tenecteplase thrombolysis for stroke up to 24 hours after onset with perfusion imaging selection: the umbrella phase IIa CHABLIS-T randomised clinical trial. Stroke Vasc Neurol. 2024 Nov 5;9(5):551-559. doi: 10.1136/svn-2023-002820. PMID 38286484